CLINICAL TRIAL: NCT04710628
Title: A Multicentric, Open-Label, Single Arm Phase II Study To Evaluate The Efficacy And Safety Of The Combination Of PEmbrolizumab And Lenvatinib In Pre-Treated Thymic Carcinoma PaTIents. PECATI.
Brief Title: Combination of Pembrolizumab and Lenvatinib, in Pre-treated Thymic CArcinoma paTIents
Acronym: PECATI
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MedSIR (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MedOPP341
Record Dates: First submitted 2020-12-03; First posted 2021-01-15 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Thymic Carcinoma; Thymoma Type B3
MeSH Terms: conditions — Thymoma | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PEMBROLIZUMAB + LENVATINIB (Experimental): Pembrolizumab 200 mg will be administered to patients as 30-minute IV infusion every 3 weeks (a window of -5 minutes and +10 minutes is permitted).
  Lenvatinib 20 mg (2 capsules of 10 mg) will be administered daily at the same time, with or without food. At the day 1 of each cycle, lenvatinib will be administered within 4 hours after finishing pembrolizumab (lenvatinib after pembrolizumab). Lenvatinib cannot be chewed
  Interventions: Drug: Pembrolizumab; Drug: Lenvatinib 10 mg

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg will be administered to patients as 30-minute intravenous infusion (a window of -5 minutes and +10 minutes is permitted) every 3 weeks.
  Other Names: MK-3475, lambrolizumab
Drug: Lenvatinib 10 mg — Lenvatinib 20 mg (2 capsules of 10 mg) will be administered daily at the same time, with or without food. At the day 1 of each cycle, lenvatinib will be administered within 4 hours after finishing pembrolizumab (lenvatinib after pembrolizumab)
  Other Names: E7080

SUMMARY:
This is a multicentric, open-label, single arm phase II study to evaluate the efficacy and safety of the combination of pembrolizumab and lenvatinib in pre-treated thymic carcinoma patients who have progressed after at least one line of platinum-based chemotherapy for advanced disease without having received any previous immunotherapy (previous bevacizumab allowed, but not sunitinib), and not amenable to curative-intent radical surgery and/or radiotherapy, regardless of PD-L1 status.

DETAILED DESCRIPTION:
Men and women aged ≥ 18 years old diagnosed with B3-thymoma or metastatic thymic carcinoma who have progressed after at least one line of platinum-based chemotherapy for advanced disease without having received any previous immunotherapy (previous bevacizumab allowed, but not sunitinib), and not amenable to curative-intent radical surgery and/or radiotherapy, regardless of PD- L1 status. Presence of measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v.)1.1 criteria. Patients are not eligible if they are candidates for a local treatment with a curative intention. Patients must present Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1 and with adequate organ function.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Relapsed / Recurrent histologically confirmed B3-Thymoma or TC patients not amenable to curative-intent radical surgery and/or radiotherapy, regardless of PD-L1 expression.
2. Patients progress after at least one previous line of platinum-based chemotherapy for advanced disease:

   a. Patients treated with neo-adjuvant or adjuvant platinum-based chemotherapy combined with radical surgery or as part of radical chemo-radiotherapy are eligible if chemotherapy was completed within 6 months before enrollment.
3. Negative result for Myasthenia Gravis (MG) by acetylcholine receptor antibodies test. Note: Acetylcholine receptor antibodies test should be performed within 6 months prior to screening visit.
4. Male/female who are at least 18 years of age on the day of signing informed consent.
5. ECOG performance status 0-1
6. Life expectancy ≥ 3 months
7. Radiological progression documented per RECIST 1.1 during or after completion of previous line therapy, per investigator's criteria.
8. Presence of measurable disease according to RECIST criteria. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.

   a. Disease status must be documented by full chest and upper abdomen (including adrenal glands) CT and/or MRI within 28 days prior study enrollment. If clinically indicated, brain imaging must be performed;
9. Provides historical (obtained archived FFPE) or fresh tumor biopsy specimen for biomarker studies, if feasible. Archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated is acceptable. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archival tissue. Note: If submitting unstained cut slides, newly cut slides should be submitted to the testing laboratory within 14 days from the date slides are cut.
10. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    1. Not a woman of childbearing potential (WOCBP) OR
    2. A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 6 months after the last dose of study treatment.
11. Has adequate bone marrow and organ function. Specimens must be collected within 10 days prior to the start of study treatment.
12. Written informed consent prior to beginning specific protocol procedures.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137).
2. Has received prior therapy with sunitinib.
3. Any evidence of active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are clinically stable (i.e. without evidence of progression by imaging for at least four weeks prior to enrollment and any neurologic symptoms have returned to baseline), and have not received steroids (for a total equivalent dose of more than 10 mg of prednisone per day) for at least 7 days prior to enrollment.
4. Uncontrolled blood pressure (Systolic BP>140 mmHg or diastolic BP >90 mmHg) in spite of an optimized regimen of antihypertensive medication.
5. Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or stroke within 6 months of the first dose of study drug, or cardiac arrhythmia requiring medical treatment at Screening.
6. Intratumor cavitation, direct invasion of main mediastinal blood vessels by the tumor or exist previous bleeding.
7. Subjects having > 1+ proteinuria on urine dipstick testing unless a 24-hour urine collection for quantitative assessment indicates that the urine protein is <1 g/24 hours.
8. Has received prior investigational agents within 4 weeks prior to allocation.
9. Participants must have recovered from all AEs due to previous therapies to ≤ Grade 1 or baseline. Participants with ≤ Grade 2 neuropathy may be eligible.
10. If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment. If surgery is needed during treatment, lenvatinib will be withheld for at least 1 week prior to elective surgery and until at least 2 weeks following major surgery and adequate wound healing. The safety of resumption of lenvatinib after resolution of wound healing has not been established.
11. Fraction ejection < 50%.
12. Known history or current evidence of active Hepatitis B (e.g., HBsAg reactive) or C (e.g., HCV RNA [qualitative] is detected) or Human Immunodeficiency Virus (HIV) (HIV-1/2 antibodies).
13. If CT has to be used, known contra-indications for CT with IV contrast.
14. Chronic use of immunosuppressive agents and/or systemic corticosteroids or any use in the last 15 days prior to enrolment:

    a. Daily prednisone at doses up to 10 mg or equivalent doses of any other corticosteroid is allowed for example as replacement therapy.
15. History of interstitial lung disease (ILD) OR pneumonitis (other than COPD exacerbation) that has required oral or IV steroids.
16. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (i.e., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
17. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.
18. Autoimmune disorders requiring immunosuppressive or dedicated treatment.
19. History of any other hematologic or primary solid tumor malignancy, unless in remission for at least 5 years and without specific treatment (as example, not allowed hormonal therapy to replace for breast cancer or hormonal therapy substitution in prostate cancer). pT1-2 prostatic cancer Gleason score < 6, superficial bladder cancer, non-melanomatous skin cancer or carcinoma in situ of the cervix are allowed.
20. Previous allogenic tissue/solid organ transplantation
21. Active infection requiring systemic therapy
22. A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

    Note: in the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.
23. Has received prior radiotherapy within 2 weeks of start of study treatment.
24. Has severe hypersensitivity (≥ Grade 3) to pembrolizumab and/or any of its excipients; known sensitivity or intolerance to lenvatinib and/or any of its excipients; severe hypersensitivity to monoclonal antibody-containing regimen.
25. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
26. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
27. Has an intestinal disease not allowing swallowing pills.
28. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through the 6 months after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 5 months
  PFS rate at 5 months, defined as the percentage of patients with B3-Thymoma and Thymic Carcinoma without disease progression at 5 months after starting the treatment combination.

SECONDARY OUTCOMES:
Response rate (RR) | 5 months
  RR with the treatment combination
Maximum tumor shrinkage (MTS) | 5 months
  MTS with the treatment combination
Disease control rate (DCR) | 5 months
  DCR with the treatment combination
Duration of response (DoR) | 5 months
  DoR with the treatment combination
Overall survival (OS) | 2 years
  OS
Incidence of Grade 3 and 4 AEs and SAEs | 2 years
  Grade 3 and 4 AEs and serious adverse events (SAEs) will be assessed, according to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v.5.0), to determine the safety and tolerability of the combination.

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Remon, MD, PhD, Principal Investigator — HM-CIOCC, Hospital HM Delfos, HM Hospitales, Barcelona (Spain); Benjamin Besse, MD, PhD, Principal Investigator — Medical Oncology Department Gustave Roussy, Villejuif (France)
Locations (13):
- France (6):
  - Institut Bergonié, Bordeaux
  - Centre Oscar Lambert, Lille
  - Hôpitaux Universitaires de Marseille - Hôpital Nord, Marseille
  - Institut Curie, Paris
  - Centre Hospitalier Universitaire de Toulouse, Toulouse
  - IGR Gustave Roussy, Villejuif
- A.O.U. San Luigi Gonzaga, Orbassano, Italy
- Spain (6):
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Sant Creu i Sant Pau, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitari i Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Remon J, Bironzo P, Girard N, Bigay-Game L, Juan-Vidal O, de Castro J, Reguart N, Greillier L, Cousin S, Dansin E, Majem M, Bernabe R, Mosquera Martinez J, Diaz M, Meya A, Alcala-Lopez D, Garcia-Sanz A, Righi L, Novello S, Besse B. Lenvatinib plus pembrolizumab in pretreated metastatic B3 thymoma and thymic carcinoma (PECATI): a single-arm, phase 2 trial. Lancet Oncol. 2025 Sep;26(9):1215-1226. doi: 10.1016/S1470-2045(25)00300-6. PMID 40907517